CLINICAL TRIAL: NCT05026788
Title: Impact of COVID-19 Pandemic on Orthopaedic Practice: the COVid-19 Emergency/Elective Related Trauma (COVERT) Collaborative
Brief Title: Impact of COVID-19 Pandemic on Orthopaedic Practice
Acronym: COVERT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Principal Investigator, Kapil Sugand, Principal Investigator, Imperial College Healthcare NHS Trust
Other Study IDs: 1414607
Record Dates: First submitted 2021-08-26; First posted 2021-08-30 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Covid19; Trauma; Orthopedic Disorder; Anesthesia; Morality
MeSH Terms: conditions — COVID-19; Wounds and Injuries; Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intra-COVID lockdown: Any patients treated for orthopaedic trauma within the mandatory lockdown due to the pandemic.
  Interventions: Other: type of treatment
- Pre/post-COVID lockdown: Any patients treated for orthopaedic trauma either before or after the imposition of lockdown induced by the pandemic.
  Interventions: Other: type of treatment

INTERVENTIONS:
Other: type of treatment — pathway of management for conservative treatment, operative treatment and type of anaesthesia used

SUMMARY:
The COVERT Collaborative is led by a group of academic surgeons that is looking into the impact of the unprecedented COVID-19 pandemic on Trauma and Orthopaedic practice. This will involve both trauma and elective procedures, as well as mortality rates, operative and anaesthetic case mix. The information will help to shape service reconfiguration and enhance patient-specific treatment especially in the threat of potential subsequent waves and future pandemics.

DETAILED DESCRIPTION:
In response to the health crisis, it is the responsibility of clinicians to audit and collaborate in order to observe the impact of the pandemic on clinical practice. With the restructure of the health infrastructure, there is likely to be changes to the nature of acute referrals to Trauma and Orthopaedics, operative and anaesthetic casemix, polytrauma and open fractures as well as the role of technology to reduce viral transmission. Patient safety ought to be prioritised at all times but a national narrative is required to equip healthcare services to counter the pandemic at various time intervals post-social distancing and lockdown at 1.5, 3, 6, 12, 18 and 24 months. This will act as an audit to compare and contrast if the reconfiguration of healthcare services is abiding by the governmental, DoH, NHS, WHO, RCS and BOA (BOAST) policies and guidelines.

ELIGIBILITY:
Inclusion Criteria:

* anyone presenting with orthopaedic trauma to the Emergency Department who has been referred to the on-call Trauma and Orthopaedic team for further management.

Exclusion Criteria:

* spinal trauma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Anyone presenting with orthopaedic trauma to the Emergency Department who has been referred to the on-call Trauma and Orthopaedic team for further management.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-03-17 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Treatment | duration of study
  Non-operative vs operative management
Mortality rate | duration of study
  For patients presenting with orthopaedic trauma
Number of COVID positive patients | duration of study
  For patients presenting with orthopaedic trauma regardless of treatment pathway

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Any data will be published in academic journals

REFERENCES:
- [Result] Park C, Sugand K, Nathwani D, Bhattacharya R, Sarraf KM. Impact of the COVID-19 pandemic on orthopedic trauma workload in a London level 1 trauma center: the "golden month". Acta Orthop. 2020 Oct;91(5):556-561. doi: 10.1080/17453674.2020.1783621. Epub 2020 Jun 23. PMID 32573331